CLINICAL TRIAL: NCT02598336
Title: Validation of Structured Light Plethysmography Against Spirometry in Children and Adults
Brief Title: Validation of Structured Light Plethysmography
Acronym: SLPvsPNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pneumacare Ltd (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP01/0010
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Disease
Keywords: Structured Light Plethysmography; Spirometry; Pneumotachograph
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breathing Sequence (Other): Simultaneous measurement using Structured Light Plethysmography and Pneumotachograph Spirometry during a period of tidal breathing followed by a forced respiratory manoeuvre. This sequence is repeated twice.
  Interventions: Device: Structured Light Plethysmography; Device: Pneumotachograph Spirometry
- Agreement and repeatability Breathing Sequence (Other): Simultaneous measurement using Structured Light Plethysmography and Pneumotachograph Spirometry during a period of tidal breathing. This sequence is repeated one further time at rest, and once further time after an exercise test to elevate respiratory rate.
  Interventions: Device: Structured Light Plethysmography; Device: Pneumotachograph Spirometry

INTERVENTIONS:
Device: Structured Light Plethysmography — Non contact device that uses light to record displacement of the anterior thorax and abdomen region
  Other Names: SLP
Device: Pneumotachograph Spirometry — Device that measures airflow at the mouth using a mouthpiece

SUMMARY:
Measurements of Structured Light Plethysmography (SLP) using a chest wall movement based method will be compared to those obtained by spirometry using a flow based pneumotachograph method. This study will enable validation of SLP in children and adults by allowing direct comparison of simultaneous measurements of breathing sequences using the two measurement techniques.

The investigators will also examine, in a group of normal adults, repeatability of the agreement between the two devices, and whether the agreement is affected by a change in tidal breathing parameters.

DETAILED DESCRIPTION:
Measurements using the Structured Light Plethysmography method will be compared to those obtained by spirometry using a flow based pneumotachograph.

Spirometry is the gold standard for measuring lung function in both clinical support and research roles. Modern spirometers are high precision, reliable instruments enabling a large numbers of parameters relating to lung volumes and the rate of emptying the lungs during a forced expiration to be measured. The most common and accurate method to measure the patient's forced expiration is via pneumotachograph which measures the flow of air through a mouthpiece and integrates the signal to derive the volume expired.

Structured Light Plethysmography (SLP) system that measures changes of the chest and abdominal wall movement during breathing by modelling the thorax and abdominal surface defined by a projected structured light pattern which enables a grid of virtual parts to be formed, the movement of which is recorded by digital cameras. SLP provides non-contact assessment to provide lung function data utilising structured light technologies and enhanced imaging processing.

In this study direct comparison will be made of measurements recorded simultaneously using the two measuring devices in children and adults.

To examine repeatability of the agreement between tidal breathing parameters measured by two techniques, repeated measurements will be performed in each of a group of normal adult subjects. The investigators will also examine whether the agreement is affected by a change in tidal breathing parameters. To obtain a change in tidal breathing parameters, measurements will be recorded during resting spontaneous breathing and after a period of exercise to elevate Respiratory Rate.

ELIGIBILITY:
Inclusion Criteria:

* For the patient group, any patient attending the outpatient department or the Lung Function Laboratory
* For the Healthy Normals group, any adult between 18 and 80 years with no current or previous respiratory condition.

Exclusion Criteria:

* A current cold or other viral infection
* chest surgery within 4 weeks
* Haemoptysis of unknown origin the (forced expiratory manoeuvre may aggravate the underlying condition)
* Pneumothorax
* Unstable respiratory or cardiovascular status (forced expiratory manoeuvre may worsen angina or cause changes in blood pressure) or recent myocardial infarction or pulmonary embolus
* Recent eye surgery
* Presence of an acute disease process that might interfere with test performance (e.g. Nausea, vomiting)

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) measured in Litres | 5 minutes
  The volume of air a person can exhale during a maximal forced breath
Forced Expiratory Volume in one second (FEV1) measured in litres per second | 5 minutes
  The volume of air a person can exhale in one second during a maximal forced breath
Peak Expiratory Flow (PEF) measured in litres per second | 5 minutes
  The maximal flow a person can achieve during a maximal forced breath

SECONDARY OUTCOMES:
Respiratory Waveform | 5 minutes
  Visual comparison of respiratory waveform shape and amplitude produced by pneumotachograph and SLP.
Respiratory Rate (RR) measured in seconds | 5 minutes
  Tmings derived from the Respiratory Waveforms
Inspiratory Time (tI) measured in seconds | 5 minutes
  Timings derived from the Respiratory Waveforms
Expiratory Time (tE) measured in seconds | 5 minutes
  Timings derived from the Respiratory Waveforms
Total breath time (tTot) measured in seconds | 5 minutes
  Timings derived from the Respiratory Waveforms
Inspiratory/expiratory ratio (tI/tE) expressed as a ratio | 5 minutes
  Timing ratios derived from the Respiratory Waveforms
The duty cycle (tI/tTot) expressed as a ratio | 5 minutes
  Timing ratios derived from the Respiratory Waveforms

OTHER OUTCOMES:
Inspiratory over Expiratory flow at 50 percent of tidal displacement (IE50) expressed at a ratio | 5 minutes
  Flow ratios derived from the Respiratory Waveforms

CONTACTS AND LOCATIONS:
Overall Officials: Karl Sylvester, PhD, Principal Investigator — Addenbrookes University Hospitals NHS Trust
Locations (1):
- Cambridge University Hospitals Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Stocks J, Godfrey S, Beardsmore C, Bar-Yishay E, Castile R; ERS/ATS Task Force on Standards for Infant Respiratory Function Testing. European Respiratory Society/American Thoracic Society. Plethysmographic measurements of lung volume and airway resistance. ERS/ATS Task Force on Standards for Infant Respiratory Function Testing. European Respiratory Society/ American Thoracic Society. Eur Respir J. 2001 Feb;17(2):302-12. doi: 10.1183/09031936.01.17203020. PMID 11334135
- [Background] Bates JH, Schmalisch G, Filbrun D, Stocks J. Tidal breath analysis for infant pulmonary function testing. ERS/ATS Task Force on Standards for Infant Respiratory Function Testing. European Respiratory Society/American Thoracic Society. Eur Respir J. 2000 Dec;16(6):1180-92. doi: 10.1034/j.1399-3003.2000.16f26.x. PMID 11292125
- [Background] Ferrigno G, Carnevali P, Aliverti A, Molteni F, Beulcke G, Pedotti A. Three-dimensional optical analysis of chest wall motion. J Appl Physiol (1985). 1994 Sep;77(3):1224-31. doi: 10.1152/jappl.1994.77.3.1224. PMID 7836125
- [Background] Cala SJ, Kenyon CM, Ferrigno G, Carnevali P, Aliverti A, Pedotti A, Macklem PT, Rochester DF. Chest wall and lung volume estimation by optical reflectance motion analysis. J Appl Physiol (1985). 1996 Dec;81(6):2680-9. doi: 10.1152/jappl.1996.81.6.2680. PMID 9018522